CLINICAL TRIAL: NCT02191241
Title: An Open, Uncontrolled Trial in Healthy Volunteers to Explore the Plasma and Urinary Pharmacokinetics of a Single Oral Dose of 1,800 mg Red Vine Leaf Extract (Antistax®)
Brief Title: Pharmacokinetics of a Single Oral Dose of 1,800 mg Red Vine Leaf Extract (Antistax®)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 1138.9
Record Dates: First submitted 2014-07-15; First posted 2014-07-16 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Healthy

ARMS (1):
- Red Vine Leaf Extract (Experimental)
  Interventions: Drug: Red Vine Leaf Extract

INTERVENTIONS:
Drug: Red Vine Leaf Extract

SUMMARY:
To describe the plasma and urinary pharmacokinetics of quercetin glucuronide and kaempferol glucuronide after the administration of a single peroral dose of 1,800mg Red Vine Leaf Extract (Antistax®). Additionally, the trial evaluated the safety and tolerability of this dose in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* male or female (if female: either of non-childbearing potential or taking adequate contraceptive measures)
* caucasian
* age: 18 to 40 years old
* body mass index (BMI): 18-28 kg x m-2
* subjects who - on the basis of extensive pre-trial investigation - could be considered to be healthy
* subjects who were willing and capable to confirm written consent to enrolment after ample information has been provided

Exclusion Criteria:

* if female: positive pregnancy test upon recruitment
* subjects with any relevant clinical abnormality (as based on extensive medical history, physical examination, vital signs)
* subjects with chronic or relevant acute infections
* subjects with therapy-requiring allergies (including drug allergies)
* subjects with suspicion of hypersensitivity to the investigational medication
* subjects with any clinically relevant laboratory abnormality (including positive results for hepatitis and HIV serology)
* subjects who had received any medication within 1 week prior to trial start or during the trial, except for hormonal contraceptives (females) or thyroid hormone replacement after thyroidectomy
* subjects who had taken a drug with a long half-life (≥ 24 hours) within one month before enrolment in the trial
* subjects who participated in a trial with a novel investigational medication within the last 8 weeks before the start of the present trial
* subjects who participated in a trial with a registered compound within the last 4 weeks before the start of the present trial
* subjects who donated blood or plasma within the last 4 weeks before the start of the present trial
* subjects who smoked more than 15 cigarettes per day and subjects who were not willing or able to abstain from smoking from 12:00 hours before and during the profiling days
* subjects known or suspected to be (social) drug dependent, incl. those drinking more than 60 g alcohol per day and who were not willing to abstain from alcohol during the active trial phase
* subjects adhering to a diet (i.e. vegetarian) or lifestyle (including extreme physical activities such as competitive sports and weight lifting) that might interfere with the investigation
* subjects known or suspected not to comply with the trial directives and/or known or suspected not to be reliable or trustworthy
* subjects known or suspected not to be capable of understanding and evaluating the information that is given to them as part of the formal information policy (informed consent), in particular regarding the risks and discomfort to which they would agree to be exposed

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2001-08; Primary Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
maximum concentration of the analyte (Cmax) | up to 24 hours after drug administration
area under the curve (AUC) extrapolated to infinity (AUC0-inf) | up to 24 hours after drug administration

SECONDARY OUTCOMES:
time to Cmax (Tmax) | up to 24 hours after drug administration
AUC under the time course of the quantifiable concentrations (AUC0-tz) | up to 24 hours after drug administration
apparent terminal disposition rate constant (λz) | up to 24 hours after drug administration
apparent terminal half-life (t1/2) | up to 24 hours after drug administration
Mean residence time (MRT) | up to 24 hours after drug administration